CLINICAL TRIAL: NCT01585545
Title: Radiomic Assessment in NSCLC: Correlation Between Multiparametric Imaging Biomarkers and Genetic Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yun Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: 2012-03-068
Record Dates: First submitted 2012-04-21; First posted 2012-04-26 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
Keywords: CT; PET CT; MRI; cancer genomics; Radiomics; Radiogenomics
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung cance tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with NSCLC

SUMMARY:
The purpose of this study is to evaluate relationships between multiparametric imaging biomarkers and genetic analysis in NSCLC patients.

DETAILED DESCRIPTION:
To evaluate relationships between multiparametric imaging biomarkers(CT, PET/CT, MRI) and genetic analysis in NSCLC patients

ELIGIBILITY:
Inclusion Criteria:

* Suspected lung cancer on chest CT or histologically proven NSCLC
* Participant is being considered for the conventional/neoadjuvant/targeted chemotherapy or surgery
* At least one measurable primary or other intrathoracic lesion >= 2cm, according to RECIST
* Performance status of 0 to 2 on the ECOG scale
* Age 20 years or older
* Able to tolerable PET/CT and CT imaging required by protocol
* Able to undergo percutaneous needle biopsy before and after chemotherapy
* Able to give study-specific informed consent

Exclusion Criteria:

* Poorly controlled diabetes
* Contraindication for CT contrast agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional and genomic profiling of lung cancer | five years
  Prognostic stratification will be evaluated using following parameters:
  1. Quantitative and qualitative parameters from CT, PET, MRI
  2. Genomic data of lung cancer samples

SECONDARY OUTCOMES:
Relationship between genomic and multiparametric imaging profiling | five years
  We will evaluate if certain relationship exists between changes in multiparametric imaging markers from CT, PET, MRI and genomic informations of NSCLC.
Precise prediction of pulmonary function such as ventilation and perfusion after the lung resection. | five years
  following parameters exracted from whole lung will be evaluated: Quantitative parameters related to pulmonary function from CT, PET, MRI 2. Prediction of longitudinal changes of pulmonary function after the lung resection

CONTACTS AND LOCATIONS:
Overall Officials: Ho Yun Lee, Dr, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea